CLINICAL TRIAL: NCT01341899
Title: Prospective Study of Autologous Hematopoietic Stem Cell Transplantation to Treat New Onset Type 1 Diabetes
Brief Title: Efficacy and Safety Study of Autologous Hematopoietic Stem Cell Transplantation to Treat New Onset Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZKX07012
Record Dates: First submitted 2011-04-21; First posted 2011-04-26 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; stem cell; C-peptide; Immune function
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Immunosuppression Therapy; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell transplantation (Experimental)
  Interventions: Procedure: immunosuppression and stem cell transplantation

INTERVENTIONS:
Procedure: immunosuppression and stem cell transplantation — Hematopoietic stem cells were mobilized with cyclophosphamide (CY, 2.0 g/m2) and granulocyte colonystimulating factor (10 μg/kg per day) and then collected from peripheral blood by leukapheresis and cryopreserved. The cells were infused after conditioning with CY (200 mg/kg) and rabbit antithymocyte globulin (4.5 mg/kg).
  Other Names: nonmyeloablative stem cell transplantation

SUMMARY:
Type 1 diabetes is an autoimmune disease and results from T cell autoimmunity mediated destruction of the majority of insulin-producing pancreatic β-cells. Hence,the development of new therapies to control T cell autoimmunity, and to preserve the remaining β-cell function will be of great significance in managing patients with type 1 diabetes

Autologous nonmyeloablative hematopoietic stem cell transplantation (AHST) has been tested for the treatment of patients with new onset of type 1 diabetes. This therapeutic strategy can result in exogenous insulin independence by destroying pathogenic memory T cells and preserving the remaining β-cell function.

However, little is known about the efficacy of AHST in the dynamics of immunocompetent cell reconstitution and how the reconstituted immune system regulates β-cell specific antibody response. Furthermore, many Chinese patients at diagnosis of type 1 diabetes have progressed to develop diabetic ketoacidosis (DKA). Whether treatment with AHST could still achieve adequate glycemic control and preserve the β-cell function and what the factors are associated with the therapeutic efficacy have not been explored.

This is a phase Ⅱ clinical trial in patients who have been diagnosed with type 1 diabetes within the previous 12 months.This study is to determine:

* The effects of autologous hematopoietic stem cell transplantation on the reconstitution of immune system
* β-cell preservation following stem cell transplantation
* The potential factors affecting efficacy of stem cell transplantation
* Whether this new therapy is safe.

DETAILED DESCRIPTION:
Patients diagnosed with type 1 diabetes within the previous 12 months will be recruited into this study.Hematopoietic stem cells were mobilized with cyclophosphamide (CY, 2.0g/m2) and granulocyte colony stimulating factor (10 μg/kg per day) and then collected from peripheral blood by leukapheresis and cryopreserved. The cells were infused after conditioning with CY (200 mg/kg) and rabbit antithymocyte globulin (4.5 mg/kg). All the included patients undergoing AHST complied with blood glucose self-monitoring and scheduled medical appointments.Their blood samples were obtained for measuring the frequency of lymphocytes and the levels of plasma hemoglobin A1c (HbA1c), serum C-peptide, islet antibodies, and cytokines longitudinally.

Ages Eligible for Study: no more than 35 years

Genders Eligible for Study: both

Islet Autoantibodies Eligible for Study: positive for glutamic acid decarboxylase antibody (GADA), protein tyrosine phosphatase antibody (IA-2A), islet cell antibody (ICA) and/or insulin autoantibody (IAAs)

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of diabetes according to the guidelines of the World Health Organization 1999
* the duration of diabetes is no more than 12 months
* positive for for glutamic acid decarboxylase antibody (GADA), protein tyrosine phosphatase antibody (IA-2A), islet cell antibody (ICA) and/or insulin autoantibody (IAAs)

Exclusion Criteria:

* pregnancy
* mental disorders
* blood diseases
* the presence of any other severe diseases that could potentially influence the transplantation outcomes

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2006-06; Primary Completion 2012-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in C-peptide levels during standard-meal tolerance test from baseline to different time points after transplantation | 3 months, 6 months, 12 months, then yearly after transplantation, up to 10 years

SECONDARY OUTCOMES:
Changes in serum levels of HbA1c from baseline to different time points after transplantation | 3 months, 6 months, 12 months, then yearly after transplantation, up to 10 years
Temporal changes of exogenous insulin requirement from baseline to different time points after transplantation | 3 months, 6 months, 12 months, then yearly after transplantation, up to 10 years
Dynamic changes in islet antibody status from baseline to different time points after transplantation | 3 months, 6 months, 12 months, then yearly after transplantation, up to 10 years
Dynamic changes in lymphocyte immunophenotyping and cytokine profiles from baseline to different time points after transplantation | 3 months, 6 months, 12 months, then yearly after transplantation, up to 10 years
mortality and dysfunction of other endocrine glands | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, MD,PhD, Principal Investigator — the Affiliated Drum Tower Hospital of Nanjing University
Locations (1):
- at Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Li L, Shen S, Ouyang J, Hu Y, Hu L, Cui W, Zhang N, Zhuge YZ, Chen B, Xu J, Zhu D. Autologous hematopoietic stem cell transplantation modulates immunocompetent cells and improves beta-cell function in Chinese patients with new onset of type 1 diabetes. J Clin Endocrinol Metab. 2012 May;97(5):1729-36. doi: 10.1210/jc.2011-2188. Epub 2012 Mar 14. PMID 22419704